CLINICAL TRIAL: NCT04829695
Title: Efficacy and Safety of Artesunate-amodiaquine (ASAQ) and Artemether-lumefantrine (AL) for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Center Region of Cameroon
Brief Title: Efficacy and Safety of Artesunate-amodiaquine and Artemether-lumefantrine for the Treatment of Malaria in Cameroon
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Yaounde 1 (Other)
Collaborators: Biotechnology Center (BTC), University of Yaounde I, Cameroon (Unknown); National Malaria Control Program (NMCP), Cameroon (Unknown); Impact Malaria, Cameroon (Unknown); Association Camerounaise pour le Marketing Social (ACMS), Cameroon (Unknown)
Responsible Party: Principal Investigator, Professor Wilfred Fon Mbacham, Professor Wilfred Fon Mbacham, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAL001/PMI/CMR
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Falciparum Malaria
Keywords: Malaria; Plasmodium falciparum; Artesunate-amodiaquine; Artemether-lumefantrine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Eligible children for whom parent/guardian informed consent are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) in the ratio 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artesunate-amodiaquine (Arm A) (Experimental): Artesunate-amodiaquine is co-packaged as artesunate 50 mg and amodiaquine hydrochloride USP equivalent to amodiaquine base of 153.1 mg. Each child shall be given one, two or three tablets depending on the weight.
  Interventions: Drug: Artesunate-amodiaquine drug combination
- Artemether-lumefantrine (Arm B) (Active Comparator): Artemether-lumefantrine is formulated as tablets and will be provided in blister packs. Each tablet contains 20 mg artemether and 120 mg lumefantrine. Every pack has a picture showing how the drug should be given and contains two blisters for each day with one, two or three tablets depending on the weight of the child.
  Interventions: Drug: Artemether-lumefantrine drug combination

INTERVENTIONS:
Drug: Artesunate-amodiaquine drug combination — Artesunate-amodiaquine is co-packaged as artesunate 50 mg and amodiaquine hydrochloride USP equivalent to amodiaquine base of 153.1 mg. Each child shall be given one, two or three tablets depending on the weight.
  Other Names: Coarsucam
  Arms: Artesunate-amodiaquine (Arm A)
Drug: Artemether-lumefantrine drug combination — Artemether-lumefantrine is formulated as tablets and will be provided in blister packs. Each tablet contains 20 mg artemether and 120 mg lumefantrine. Every pack has a picture showing how the drug should be given and contains two blisters for each day with one, two or three tablets depending on the weight of the child.
  Other Names: Coartem
  Arms: Artemether-lumefantrine (Arm B)

SUMMARY:
Malaria remains a major public health concern in Cameroon especially among vulnerable groups such as children less than five years and pregnant women. Artesunate-amodiaquine (ASAQ) and artemether-lumefantrine (AL) have been used for the treatment of uncomplicated Plasmodium falciparum in Cameroon since 2004. Worldwide, several studies among children have reported high efficacy and safety of artemisinin-based combination therapies (ACTs). There is paucity of data to support the continuous use of ASAQ and AL in Cameroon. The main objective of this study is to assess the efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine during a 28-day follow-up period in children with acute uncomplicated P. falciparum malaria in the Center Region of Cameroon. A randomized, open-labelled, controlled clinical trial comparing artesunate-amodiaquine (ASAQ) and artemether-lumefantrine (AL) will be carried out from 5th April to 31st December, 2021 at six hospitals in the Center Region of Cameroon. The study participants shall include febrile patients aged 6 months to 10 years with confirmed uncomplicated P. falciparum infection. Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) in the ratio 1:1. A minimum sample of 76 patients will be required for the study. With a 20 % increase to allow loss to follow-up and withdrawals during the 28-day follow-up period, 92 patients will be enrolled for each of the two study arms. The study will recruit a total of 184 patients. However, since 6 sites will be involved, a minimum of 30 participants shall be enrolled per site. Drug intake will be done under strict supervision on days 0, 1 and 2. Follow-up visits will be performed on days 3, 7, 14, 21, and 28 to evaluate clinical and parasitological resolution of their malaria episode as well as adverse events. Polymerase chain reaction (PCR) genotyping of merozoite surface proteins 1 and 2 (msp-1, msp-2) as well as glutamate rich protein (GLURP) will be used to differentiate between recrudescence and new infection.

DETAILED DESCRIPTION:
Brief title: Efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine for the treatment of malaria in Cameroon.

Official title: Monitoring the efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria among children in the Center Region of Cameroon.

Purpose: To monitor the efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria among children in the Center Region of Cameroon.

Background: Malaria remains a major public health concern in Cameroon especially among vulnerable groups such as children less than 5 years and pregnant women. artesunate-amodiaquine (ASAQ) and artemether-lumefantrine (AL) are currently being used for the treatment of uncomplicated Plasmodium falciparum in Cameroon. Worldwide, several studies among children have reported high efficacy and safety of artemisinin-based combination therapies (ACTs). There is paucity of data to support the continuous use of ASAQ and AL in Cameroon.

Objective: To assess the efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine during a 28-day follow-up period among children with acute uncomplicated P. falciparum malaria in Center Region of Cameroon.

Study sites: District Hospital Akonolinga, District Hospital Mfou, District Hospital Soa, District Hospital Mbalmayo, District Hospital Mbandjock, and District Hospital Ngog-Mapubi in the Center Region of Cameroon.

Study period: 5th April to 31st December, 2021. Study design: This surveillance study is a two arm, open label, randomized controlled clinical trial.

Patient population: Febrile patients aged 6 months to 10 years, with confirmed uncomplicated P. falciparum infection. Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) in the ratio 1:1.

Sample size: A minimum sample of 76 patients will be required for the study. With a 20 % increase to allow loss to follow-up and withdrawals during the 28-day follow-up period, 92 patients will be enrolled for each of the two study arms. The study will recruit a total of 184 patients. At least 30 participants shall be enrolled at each of the six study sites.

Treatment (s) and follow-up: Drug intake will be done under strict supervision on days 0, 1 and 2. Follow-up visits will be performed on days 3, 7, 14, 21, and 28 to evaluate clinical and parasitological resolution of their malaria episode as well as adverse events. Polymerase chain reaction (PCR) genotyping of merozoite surface proteins 1 and 2 (msp-1, msp-2) as well as glutamate rich protein (GLURP) will be used to differentiate between recrudescence and new infection.

Classification of treatment outcomes: Classification of treatment outcomes will be done based on the WHO 2009 guidelines: treatment failure (Early Treatment Failure-ETF, Late Clinical failure-LCF and Late Parasitological Failure-LPF) and treatment success (Adequate Clinical and Parasitological Response-ACPR).

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender, aged 6 months to 10 years will be recruited.
* Uncomplicated P. falciparum malaria confirmed by microscopy using Giemsa-stained thick film with an asexual parasite density within the range 1000 to 200000 parasites/μl.
* Presenting with fever (axillary temperature ≥ 37.5oC) or having a history of fever in the preceding 24 hours.
* Able to ingest tablets orally (either suspended in water or uncrushed with food).
* Willing to participate in the study with written informed consent from parent/guardian.
* Willing and able to attend the clinic on stipulated regular follow-up visits.

Exclusion Criteria:

* Mixed or mono-infection with another Plasmodium species detected by microscopy.
* Children who are currently suffering or had the following within the last 2 months: tuberculosis, HIV, schistosomiasis, diabetes mellitus, cardiovascular disease, gout, rheumatoid arthritis, underlying chronic hepatic or renal disease, hypoglycaemia, jaundice, respiratory distress, and other inflammatory-related diseases.
* Signs/symptoms indicating severe/complicated malaria" according to WHO criteria (WHO definition) such as:

  1. Not able to drink or breastfeed.
  2. Persistent vomiting (>2 episodes within the previous 24 hours).
  3. Convulsions (>1 episode within the previous 24 hours).
  4. Lethargic/unconscious.
  5. Severe anemia (hemoglobin < 5 g/dl).
* Serious gastrointestinal disease.
* Presence of severe malnutrition defined as a child aged between 6-60 months whose weight-for-height is below -3 z-score (W/H < 70%) or has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 115 mm).
* Regular medication, which may interfere with anti-malarial pharmacokinetics.
* History of hypersensitivity reactions or contraindications to any of the medicine (s) being tested or used as alternative treatment (s).
* Individuals who have taken part in anti-malarial efficacy and safety studies in the last 3 months.
* Participants who have taken anti-malarial drugs within the last one month.

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2021-04-05 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment success and adverse events following treatment with ASAQ and AL during 28 days follow-up period in children with uncomplicated P. falciparum malaria | 10 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) and follow-up will be done for a duration of 28 days.

SECONDARY OUTCOMES:
Proportion of patients with early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response as indicators of efficacy according to the WHO 2009 guidelines | 10 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) and follow-up will be done for a duration of 28 days. Recrudescence will be distinguished from re-infection by polymerase chain reaction (PCR) analysis.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 10 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) and follow-up will be done for a duration of 28 days.
Number of children with single nucleotide polymorphisms of P. falciparum genes responsible for resistance to ASAQ and AL | 10 months
  Pre-treatment and recrudescence/reinfection samples during follow-up shall be used to characterize the molecular markers of Plasmodium falciparum chloroquine resistant transporter(Pfcrt), Plasmodium falciparum multi-drug resistant 1 (Pfmdr1), and Plasmodium falciparum K13 (Pfk13) propellar domain conferring resistance to artemisinins or partner drugs.
Number of children with single nucleotide polymorphisms of P. falciparum histidine-rich protein 2 and 3 genes | 10 months
  Pre-treatment shall be used to detect single nucleotide polymorphisms present in Plasmodium falciparum histidine-rich protein 2 and 3 genes.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Fon Mbacham, PhD, Principal Investigator — University of Yaounde I

IPD SHARING:
Plan to Share IPD: Yes
Research findings will be communicated with the scientific community and policymakers. This will be done through public engagements and publications in peer-review journals.
Supporting Information: Study Protocol, CSR
Time Frame: 31st December 2021 for at least 10 years
Access Criteria: Not available for now